CLINICAL TRIAL: NCT03849326
Title: Chronic Fatigue Etiology in Intensive Care Unit Survivors: the Role of Neuromuscular Function
Acronym: FatPostRéa
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to the health crisis and the lack of staff in the department no inclusion could be realized
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: University of Saint-Etienne (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 18CH175; 2018-A03511-54 (Other: ANSM)
Record Dates: First submitted 2019-02-19; First posted 2019-02-21 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Chronic Fatigue Syndrome; Intensive Care Unit; Muscle
Keywords: Neuromuscular function
MeSH Terms: conditions — Fatigue Syndrome, Chronic | interventions — Surveys and Questionnaires; Hematologic Tests; Actigraphy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Non-fatigued" patients (Experimental)
  Interventions: Other: Questionnaires; Biological: blood test; Other: Maximal effort test; Device: actigraphy; Device: Neuromuscular evaluation
- "Fatigued" patients (Experimental)
  Interventions: Other: Questionnaires; Biological: blood test; Other: Maximal effort test; Device: actigraphy; Device: Neuromuscular evaluation

INTERVENTIONS:
Other: Questionnaires — Quality of life Depression Physical pain Social provisions Quality of sleep
Biological: blood test — complete blood count and cytokine concentration
Other: Maximal effort test — The maximal effort test with VO2max recordings will be assessed during the first visit to the laboratory.
Device: actigraphy — assessment of sleep quality
Device: Neuromuscular evaluation — * The maximum isometric force produced by the knee extensors will be measured on the ergometer
  * the intensity of muscular electrical activity recorded by surface electromyography
  * Peripheral nerve stimulation
  * Transcranial magnetic stimulation
  * Magnetic resonance imaging (optional)

SUMMARY:
Chronic fatigue is the most common and debilitating symptom in intensive care unit (ICU) survivors. Indeed, it has been widely reported that patients who stayed in ICU for prolonged periods report a feeling of tiredness for months to years after ICU discharge. This chronic fatigue affects their quality of life by decreasing their capacity to perform simple tasks of daily life.

The aim of the present project is to determine whether deteriorated neuromuscular function (i.e. increased fatigability) is involved in this feeling of chronic fatigue. Because the causes of this feeling are multi-dimensional, a large battery of tests will allow us to better understand the origin of chronic fatigue. A better knowledge of chronic fatigue etiology will allow to optimize rehabilitation treatments to decrease the apparition/persistence of chronic fatigue and in fine improve life quality.

ELIGIBILITY:
Inclusion Criteria:

* Have been ventilated for at least 72 hours in the intensive care unit
* IGS2 score (severity in resuscitation) > 15
* FACIT-F (Functional Assessment of Chronic Illness Therapy-Fatigue) score ≥ 36 or a score ≤ 32
* intensive care unit discharge in ≥ 6 months and ≤ 5 years preceding the study
* Approval received from a physician
* Command of the French language

Exclusion Criteria:

* Taking neuroactive substances that can alter corticospinal excitability
* Contraindication to the application of a magnetic field
* Contraindication to the practice of Magnetic Resonance Imaging
* Participant is pregnant
* Patients with psychiatric disorders
* Paraplegic and hemiplegic patients
* Addictive disorders

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-12 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
voluntary maximum force reduction | at 2 weeks

SECONDARY OUTCOMES:
Neuromuscular function : cortical activity | at 2 weeks
  Level of cortical activation and cortico-spinal excitability measured by transcranial magnetic stimulation
Neuromuscular function : Peripheral function | at visit 2
  Peripheral function by electrical nerve stimulation
Maximal oxygen uptake (VO2max) | at 2 weeks
  measured by effort test
quality of sleep | at baseline
  measured by actigraphy
Quadriceps muscle volume (optional) | at 3 weeks
  with Magnetic resonance imaging
muscle dysfunction (optional) | at 3 weeks
  measured by a Phosphorus 31 Nuclear magnetic resonance test

CONTACTS AND LOCATIONS:
Overall Officials: Jérome MOREL, MD PhD, Principal Investigator — CHU de Saint Etienne
Locations (1):
- Hôpital privé de la Loire, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No